CLINICAL TRIAL: NCT00522301
Title: A Phase II Trial of Oral Sorafenib (Bay43-9006) In Women With Epithelial Ovarian, Fallopian Tube Or Peritoneal Carcinoma In Second Or Greater Remission
Brief Title: Sorafenib in Treating Patients With Ovarian Epithelial Cancer, Fallopian Tube Cancer, or Peritoneal Cancer in at Least the Second Remission
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-080; P30CA008748 (NIH); MSKCC-07080; BAYER-MSKCC-07-080
Record Dates: First submitted 2007-08-28; First posted 2007-08-29 (Estimated); Results first posted 2016-02-29 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; fallopian tube cancer; primary peritoneal cavity cancer; stage I ovarian epithelial cancer; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Sorafenib; Immunoenzyme Techniques; Immunohistochemistry

ARMS (1):
- Oral Sorafenib (BAY43-9006) (Experimental): Sorafenib is supplied as 200-mg tablets. Sorafenib will be administered as 400 mg orally daily x 28 days (continuous). One cycle = 28 days. There is no planned treatment interruption between cycles. Sorafenib should be taken without food (at least 1 hour before or 2 hours after eating). In the absence of intolerable toxicity, a patient may continue to receive treatment with sorafenib until disease progression, or until 24 months have elapsed.
  Interventions: Drug: sorafenib tosylate; Other: immunoenzyme technique; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: sorafenib tosylate
Other: immunoenzyme technique
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Other: pharmacological study

SUMMARY:
RATIONALE: Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well sorafenib works in treating patients with ovarian epithelial cancer, fallopian tube cancer, or peritoneal cancer in at least the second remission.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the 12-month progression-free survival (PFS) rate of women with ovarian epithelial, fallopian tube, or peritoneal cancer in second or greater remission treated with oral sorafenib tosylate.

Secondary

* To determine the safety and tolerability of prolonged treatment with oral sorafenib tosylate in women with a history of recurrent ovarian cancer.
* To correlate serum markers of angiogenesis (i.e., VEGF and bFGF) and tumor markers pAKT, HIF-1 α , and VEGF with 12-month PFS.

OUTLINE: Patients receive oral sorafenib twice a day on days 1-28. Treatment repeats every 28 days for up to 24 months in the absence of disease progression or unacceptable toxicity.

Patients undergo tumor tissue and blood sample collection at baseline, every 12 weeks during study, and after completion of study therapy for pharmacokinetic studies. Samples are analyzed for soluble markers of angiogenesis (i.e., VEGF and bFGF) via ELISA and HIF-1 α, VEGF, and pAKT via IHC staining.

After completion of study treatment, patients are followed at 4 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed epithelial carcinoma arising in the ovary, fallopian tube, or peritoneum

  * Any stage and grade at diagnosis
* Must have received initial cytoreductive surgery and chemotherapy with ≥ 1 platinum-based chemotherapy regimen

  * Persistent or recurrent disease after initial therapy
* In complete clinical remission after chemotherapy for recurrent disease, meeting all of the following criteria:

  * CA125 ≤ 35 units/L
  * Normal physical examination
  * No definite evidence of disease by CT scan of the abdomen and pelvis

    * Lymph nodes and/or soft tissue abnormalities ≤ 1.0 cm are not considered definite evidence of disease
* No known brain metastases

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Karnofsky performance status 70-100%
* Life expectancy > 3 months
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9.0 g/dL
* INR < 1.5 OR PT/PTT within normal limits
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Urinalysis negative for protein

  * If urinalysis shows 1+ protein by dipstick or protein ≥ 30-100 mg/dL by semi-quantitative assay, a 24-hour urine collection is required

    * Eligible patients must have a total urinary protein ≤ 500 mg AND measured creatinine clearance ≥ 50 mL/min from a 24-hour urine collection
* Bilirubin ≤ 1.5 times ULN
* AST and ALT ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* Stable blood pressure (BP) measurement required on 3 separate days prior to the start of treatment
* No peripheral neuropathy > grade 1
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

Exclusion criteria:

* Other invasive malignancies within the past 5 years, except nonmelanoma skin cancer
* Uncontrolled concurrent illness or medical condition including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Uncontrolled diabetes
* Psychiatric illness or social situation that would preclude study compliance
* Uncontrolled hypertension defined as a persistent BP > 150/100 mm Hg (or a persistent BP > 180/90 mm Hg if the patient has a history of isolated systolic hypertension) despite ≥ 2 attempts at antihypertensive medication dosage adjustment ≥ 2 weeks apart
* Thrombolic or embolic events such as cerebrovascular accident, including transient ischemic attack, within the past 6 months
* Pulmonary hemorrhage or bleeding event ≥ grade 2 within 4 weeks of the first dose of study drug
* Other hemorrhage or bleeding event ≥ grade 3 within 4 weeks of the first dose of study drug
* Serious nonhealing wound, ulcer, or bone fracture
* Evidence or history of bleeding diathesis or coagulopathy
* Inability to take oral medications or gastrointestinal condition that compromises absorption
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to sorafenib tosylate

PRIOR CONCURRENT THERAPY:

Inclusion criteria:

* See Disease Characteristics
* No prior sorafenib tosylate or other inhibitors of MAPK signaling intermediates or angiogenesis inhibitors
* No prior cancer treatment that would contraindicate protocol therapy
* More than 4 weeks since prior radiotherapy
* More than 3 weeks since prior chemotherapy, biological therapy, or immunotherapy
* More than 1 week since prior hormonal therapy for cancer treatment

Exclusion criteria:

* Major surgery (i.e., laparotomy) within the past 4 weeks or minor surgery within the past 2 weeks

  * Placement of a vascular access device is not considered minor surgery
* Concurrent combination antiretroviral therapy for HIV-positive patients
* Concurrent St. John wort, rifampin, or enzyme-inducing anticonvulsants (e.g., carbamazepine, phenytoin, or phenobarbital)

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-07; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William P. Tew, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Paul Sabbatini, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan - Kettering Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral Sorafenib (BAY43-9006): Sorafenib will be administered as 400 mg orally daily x 28 days (continuous).
Period: Overall Study
Arm/Group | Oral Sorafenib (BAY43-9006)
Started | 6
Completed | 0
Not Completed | 6
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 5

BASELINE CHARACTERISTICS:
Arm/Group | Oral Sorafenib (BAY43-9006)
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Rate at 12 Months
Description: All 5 patients experienced a rash. As a result, all 5 were either advised to withdraw from the protocol, or withdrew themselves from the protocol. The outcome was not met.
Time Frame: 1 year
Population: Protocol terminated prior to primary outcome evaluation. All 5 patient were evaluable for toxicity only.
Arm/Group | Oral Sorafenib (BAY43-9006)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Oral Sorafenib (BAY43-9006)
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Sorafenib (BAY43-9006) (N=5)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Sorafenib (BAY43-9006) (N=5)
Rash (Skin and subcutaneous tissue disorders) | 5 (5)
Dizziness (Nervous system disorders) | 5 (5)
Pain (General disorders) | 2 (2)
Fatigue (General disorders) | 5 (5)
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 5 (5)
Alkaline Phosphatase (Metabolism and nutrition disorders) | 5 (5)

LIMITATIONS AND CAVEATS:
Early termination as it would not meet it's primary endpoint of improved survival. None of the patients completed the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes